CLINICAL TRIAL: NCT07395752
Title: Development and Biological Efficacy Validation of Youth Suicide and Self-Harm Intervention Program
Brief Title: Youth Suicide and Self-Harm Intervention: Clinical and Biological Outcomes Study
Acronym: SHIELD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Sungshin Women's University (Other)
Responsible Party: Principal Investigator, Yunmi Shin, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS-2024-00409433
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Suicidal Ideation; Self-Injurious Behavior; Suicide, Attempted
Keywords: Youth suicide; Suicidal ideation; Suicide attempt; fMRI; Social rhythm; Adolescents; Young adults
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior; Suicide, Attempted | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the intervention program or a usual-care comparison group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participant assignment to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Youth Suicide and Self-Harm Intervention Program (Experimental): A structured modular intervention program integrating mindfulness-based techniques, Dialectical Behavior Therapy (DBT) skills, and social rhythm stabilization strategies for adolescents and young adults at elevated risk for suicide and self-harm.
  The program includes tailored modules addressing:
  suicidal ideation and self-injurious thoughts/behaviors emotion regulation and distress tolerance (DBT-informed) mindfulness and attention regulation sleep and social rhythm stabilization crisis response and safety planning
  Modules are delivered by trained clinicians using a standardized manual, with components adjusted to the developmental needs of adolescents versus young adults. Participants complete psychological and biological assessments (e.g., resting-state fMRI) at baseline and follow-up.
  Interventions: Behavioral: Self-Harm Intervention and Education for Long-term Development (SHIELD) Program
- General Mental Health Education Program (Active Comparator): Participants in the active comparator group will receive a general mental health education program of equal duration and session frequency as the intervention group.
  The education program covers topics such as:
  understanding stress and mood
  healthy coping strategies
  lifestyle factors related to mental well-being
  sleep hygiene
  healthy routines and social relationships
  This program does not include suicide- or self-harm-specific therapeutic components, nor modular DBT/mindfulness/rhythm stabilization strategies used in the intervention group.
  Participants complete the same baseline and follow-up psychological and biological assessments as the intervention group.
  Interventions: Behavioral: General Mental Health Education

INTERVENTIONS:
Behavioral: Self-Harm Intervention and Education for Long-term Development (SHIELD) Program — A structured, module-based psychological intervention program consisting of 8 weekly sessions. The program is tailored into three customized tracks based on the participant's age and clinical needs:
  * Common Core Module (Cross-cutting): Social Rhythm Therapy (SRT) is applied to all participants starting from Session 2 to stabilize daily routines (sleep, meals, activities) and reduce emotional impulsivity.
  * Track 1: Youth Self-Harm Program (Ages 14-18): Focuses on functional understanding of non-suicidal self-injury, mindfulness-based emotion regulation, interpersonal skills, and behavioral therapy.
  * Track 2: Youth Suicide Program (Ages 14-18): Includes an intensive behavioral therapy session (Session 3) for crisis analysis, followed by mindfulness, interpersonal skills, and cognitive therapy modules to enhance resilience and prevent suicide attempts.
  * Track 3: Young Adult Program (Ages 19-30): Addresses both self-harm and suicide-related issues through personalized modules inc
  Arms: Youth Suicide and Self-Harm Intervention Program
Behavioral: General Mental Health Education — Participants watch 8 educational videos over an 8-week period. The education is ideally conducted at the research site. Similar to the intervention group, participants are also required to use a wearable device during the study period.
  Arms: General Mental Health Education Program

SUMMARY:
The goal of this clinical trial is to develop and evaluate youth-focused intervention programs for suicide and self-harm that are tailored to the psychological, developmental, and cultural characteristics of Korean adolescents and young adults. The study examines whether two structured, mindfulness-based intervention programs-one for middle and high school students and one for young adults-reduce suicidal ideation, self-harm behaviors, depressive symptoms, and emotion-regulation difficulties.

The study also aims to determine whether these clinical improvements are associated with biological changes, including alterations in resting-state functional brain activity (e.g., ALFF, ReHo, and functional connectivity) and social rhythm patterns.

The main questions this study seeks to answer are:

* Does the youth suicide and self-harm intervention program reduce suicidal ideation and self-injurious thoughts/behaviors?
* Does the program improve mood, sleep, hopelessness, and emotion regulation?
* Are improvements in clinical outcomes accompanied by changes in biological markers of suicide risk?
* Researchers will compare the intervention program to usual care provided in hospitals, schools, and community mental health settings.

Participants will:

* Participate in the structured suicide/self-harm intervention program or receive usual care.
* Complete standardized assessments of mood, sleep, emotion regulation and suicide/self-harm risk.
* Undergo biological assessments, including resting-state fMRI and rhythm-related measures, at baseline and follow-up.
* Be followed for up to 12 weeks.

DETAILED DESCRIPTION:
This study is part of a national research initiative aimed at addressing youth suicide and self-harm, which have shown persistent increases and earlier onset in Korea. Despite the existence of many prevention programs, their effectiveness has been limited due to insufficient implementation strategies, lack of biological evidence, and the absence of structured, field-ready manuals or expert training systems. To overcome these limitations, this project seeks to develop, validate, and disseminate comprehensive suicide and self-harm intervention programs for adolescents and young adults.

The study develops two tailored intervention programs-one for middle and high school students and one for young adults-based on mindfulness-informed and evidence-based techniques. The intervention differentiates between suicide and non-suicidal self-injury, addressing each with distinct therapeutic modules that reflect their unique psychological and neurobiological mechanisms. The programs will include emotion regulation skills, crisis response strategies, behavioral techniques, and structured manuals for both therapists and participants.

Alongside the intervention, the study develops the first Korean clinical practice guidelines (CPGs) for suicide and self-harm in adolescents and young adults, based on extensive literature review, international guideline comparison, and expert consensus.

The effectiveness of the intervention will be tested using a randomized or quasi-experimental design across multiple settings, including hospitals, community mental health centers, and schools. Clinical outcomes include suicidal ideation, self-harm behaviors, depressive symptoms, hopelessness, sleep disturbance, emotion regulation, and social rhythm stability. Biological outcomes will be evaluated using resting-state fMRI metrics (ALFF, ReHo, and functional connectivity) and other physiological indicators that reflect neural circuits implicated in suicide risk.

The goal is to establish both clinical and biological evidence for the effectiveness of the program, achieve national certification for two intervention programs and one training curriculum, and ultimately develop an implementation model that can be scaled across community and clinical settings in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. General Criteria

   * Aged between 15 and 30 years
   * Obtained informed consent from a parent or legal guardian for participants under 19 years of age
2. For the Self-Harm Group

   * At least one incident of non-suicidal self-injury (NSSI) within the last 6 months
   * Self-Harm Screening Inventory (SHSI) score of at least 1 (at least one "Yes" response)
3. For the Suicide Attempt Group

   * Suicide attempt within the last 6 months
   * Depressive Symptom Inventory-Suicidality Subscale (DSI-SS) score of 3 or higher

Exclusion Criteria:

1. Psychiatric and Developmental Conditions

   * History of developmental disorders, including intellectual disability or autism spectrum disorder
   * Diagnosis of schizophrenia or bipolar disorder
   * Currently in an acute psychotic state
2. Medical and Physical Conditions

   * Presence of severe physical illness that interferes with daily life
   * Presence of metallic substances in the body (e.g., cardiac pacemakers, artificial heart valves) that are incompatible with fMRI
   * Diagnosis of claustrophobia
   * Current Treatment and Intervention
   * Currently receiving regular and active cognitive behavioral therapy (CBT)
   * Initiation of pharmacological treatment within the last 2 months
3. Communication and Consent

   * Inability to communicate fluently in Korean
   * Failure to obtain informed consent from a parent or legal guardian for participants under 19 years of age

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Suicidality (DSI-SS Score) | Baseline and Week 8, Baseline and Week 12
  The DSI-SS is a 4-item self-report questionnaire designed to assess the frequency and intensity of suicidal ideation and impulses. Scores range from 0 to 12, with higher scores indicating greater severity of suicidality; a score of 3 or higher is considered the clinical cut-off for high suicide risk.
Change from Baseline in Functional Assessment of Self-Mutilation (FASM) Frequency Score | Baseline and Week 8, Baseline and Week 12
  The FASM assesses the methods and frequency of non-suicidal self-injury (NSSI), as well as the functions maintaining the behavior. It distinguishes between Internal Functions (e.g., emotion regulation) and Social Functions (e.g., influencing others). The instrument yields data on the total frequency of self-mutilative behaviors and separate scores for these functional domains.
Change from Baseline in Self-Harm Screening Inventory (SHSI) Total Score | Baseline and Week 8, Baseline and Week 12
  The SHSI is a 10-item self-report measure used to screen for non-suicidal self-injury (NSSI) behaviors over the past year. It assesses 10 specific methods of self-harm (e.g., cutting, hitting, overdosing) performed without the intent to die. Each item is scored as 0 (No) or 1 (Yes). Total scores range from 0 to 10; a score of 1 or higher (indicating any experience of self-harm) is the cut-off for recommending a visit to a psychiatrist.
Change from Baseline in Circadian rhythm stability | Through the end of the intervention period (approximately 12 weeks)
  Circadian rhythm stability refers to the consistency of 24-hour rest-activity patterns across days, as assessed using wrist-worn actigraphy.
  Inter-daily Stability (IS) quantifies the degree of similarity between daily activity profiles across consecutive days, with values ranging from 0 to 1. Higher IS values indicate greater stability and synchronization of the circadian rest-activity rhythm.
Researcher-Defined NSSI and Suicide Attempt Frequency | Baseline and Week 8, Baseline and Week 12
  These researcher-defined items assess the frequency of Non-Suicidal Self-Injury (NSSI) and suicide attempts. NSSI frequency is measured across four timeframes (lifetime, past year, past month, past week) using a 7-point ordinal scale ranging from 'Once' to '50 times or more'. Suicide attempts are assessed by total lifetime frequency (4-point scale) and the recency of the most recent attempt. Higher scores on frequency items indicate a greater number of incidents.
Change from Baseline in Social Rhythm Stabilization | Daily throughout the intervention period (8 weeks)
  The Social Rhythm Stabilization Score assesses the regularity of daily routines (e.g., sleep, activities) through the completion of a daily social rhythm log. Variability is derived using 'Max-Min' for durations and 'Circular Time Distance' for clock times. Lower values indicate greater stability. Scores are categorized as: Very Regular (≤ 30), Regular (31-60), Mildly Variable (61-90), Variable (91-120), Irregular (121-180), and Very Irregular (> 180).

SECONDARY OUTCOMES:
Change from Baseline in Barratt Impulsiveness Scale (BIS-II) Total Score | Baseline and Week 8, Baseline and Week 12
  The BIS-II is a 23-item questionnaire designed to assess the personality construct of impulsiveness. Total scores range from 23 to 92, where higher scores indicate higher levels of impulsiveness.
Change from Baseline in Difficulties in Emotional Regulation Scale-Short Form (DERS-SF) Total Score | Baseline and Week 8, Baseline and Week 12
  The DERS-SF is an 18-item self-report measure used to assess difficulties in emotion regulation. Scores range from 18 to 90, where higher scores indicate greater difficulty in emotion regulation.
Change from Baseline in Distress Tolerance Scale (DTS) Total Score | Baseline and Week 8, Baseline and Week 12
  The DTS is a 15-item self-report measure of emotional distress tolerance. Scores range from 15 to 75, with higher scores indicating higher levels of distress tolerance (i.e., better capacity to withstand distress).
Change from Baseline in Generalized Anxiety Disorder-7 (GAD-7) Total Score | Baseline and Week 8, Baseline and Week 12
  The GAD-7 is a 7-item instrument used to assess the severity of generalized anxiety. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. Severity categories are defined as Mild (5-9), Moderate (10-14), and Severe (15-21). A total score of 10 or greater is the clinical cut-off for identifying probable generalized anxiety disorder.
Change from Baseline in Patient Health Questionnaire (PHQ-9) Total Score | Baseline and Week 8, Baseline and Week 12
  The PHQ-9 is a 9-item module used to screen for and measure the severity of depression. Scores range from 0 to 27, where higher scores indicate greater severity of depressive symptoms.
Change from Baseline in Perceived Stress Scale (PSS) Total Score | Baseline and Week 8, Baseline and Week 12
  The PSS is a 10-item instrument used to measure the perception of stress. Scores range from 0 to 40, with higher scores indicating higher levels of perceived stress. Stress levels are categorized as Low (0-13), Moderate (14-26), and High (27-40).
Change from Baseline in Ruminative Response Scale-Short Form (RRS-SF) Total Score | Baseline and Week 8, Baseline and Week 12
  The RRS-SF is a 10-item measure that assesses rumination in response to depressed mood. Scores range from 10 to 40, where higher scores indicate higher levels of rumination.
Change from Baseline in UCLA Loneliness Scale (ULS-6) Total Score | Baseline and Week 8, Baseline and Week 12
  The ULS-6 is a 6-item scale designed to measure subjective feelings of loneliness and social isolation. Scores range from 0 to 18, where higher scores indicate higher levels of loneliness.
Change from Baseline in Perceived Invalidation of Emotion Scale (PIES) Total Score | Baseline and Week 8, Baseline and Week 12
  The PIES is a 10-item instrument that measures the extent to which an individual perceives their emotions as being invalidated by others. Total scores range from 10 to 50, where higher scores indicate higher levels of perceived emotional invalidation.
Change from Baseline in Rosenberg Self-Esteem Scale (RSES) Total Score | Baseline and Week 8, Baseline and Week 12
  The RSES is a 10-item scale that measures global self-worth. Scores range from 10 to 40, with higher scores indicating higher self-esteem.
Change from Baseline in Insomnia Severity Index (ISI) Total Score | Baseline and Week 8, Baseline and Week 12
  The ISI is a 7-item instrument measuring the nature, severity, and impact of insomnia. Scores range from 0 to 28, with higher scores indicating more severe insomnia symptoms.
Change from Baseline in Pediatric Daytime Sleepiness Scale (PDSS) Total Score | Baseline and Week 8, Baseline and Week 12
  The PDSS is an 8-item self-report measure of daytime sleepiness in school-aged children. Scores range from 0 to 32, with higher scores indicating greater daytime sleepiness.
Change from Baseline in Sleep Health Index (SHI) Score | Baseline and Week 8, Baseline and Week 12
  The Sleep Health Index (SHI) is a 16-item instrument that assesses sleep health across three sub-domains: Sleep Quality, Sleep Duration, and Sleep Disorders. Raw scores are converted into a standardized index ranging from 0 to 100. A higher score indicates better sleep health.

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Medical Center, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Due to the sensitive nature of the data regarding self-harm and suicidality among vulnerable populations, IPD sharing is currently undecided to ensure participant confidentiality and ethical compliance.